CLINICAL TRIAL: NCT00985712
Title: A Randomized, Open-label Study on the Effects of Insulin Pen Devices on Glycemic Control in Children, Adolescents and Adults With Type 1 Diabetes: Novel Pen With Memory Function (HumaPen Memoir) vs. Conventional Pen Without Memory Function (HumaPen Luxura)
Brief Title: A Study on the Effect of 2 Pen Devices on HbA1c
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12704; H9D-SB-ITAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-09-23; First posted 2009-09-28 (Estimated); Results first posted 2012-06-04 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HumaPen Luxura (Experimental): Participant's insulin dose of Insulin Lispro or Huminsulin Normal is delivered subcutaneously via HumaPen Luxura daily for 24 weeks
  Interventions: Drug: Insulin Lispro; Drug: Huminsulin Regular; Device: HumaPen Luxura
- HumaPen Memoir (Experimental): Participant's insulin dose of Insulin Lispro or Huminsulin Normal is delivered subcutaneously via HumaPen Memoir daily for 24 weeks
  Interventions: Drug: Insulin Lispro; Drug: Huminsulin Regular; Device: HumaPen Memoir

INTERVENTIONS:
Drug: Insulin Lispro — subcutaneously, daily (as determined by patient's blood glucose), for 24 weeks
  Other Names: Humalog; LY275585
Drug: Huminsulin Regular — subcutaneously, daily (as determined by patient's blood glucose), for 24 weeks
  Other Names: Huminsulin Normal; LY041001
Device: HumaPen Memoir — subcutaneously, daily for 24 weeks
  Arms: HumaPen Memoir
Device: HumaPen Luxura — subcutaneously, daily for 24 weeks
  Arms: HumaPen Luxura

SUMMARY:
The purpose of this study is to test the hypothesis that the HumaPen Memoir with memory function, when used over 24 weeks for prandial insulin injections achieves superior glycemic control, when compared to the conventional HumaPen Luxura without memory function.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* receiving at least 3 prandial injections per day with short-acting or analogue insulin

Exclusion Criteria:

* Insulin pump therapy
* receiving pre-mixed insulin preparations

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (29):
- Germany (29):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aschaffenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aßlar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Mergentheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bosenheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Diez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Falkensee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flensburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fulda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giessen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herdecke
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuwied
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rehlingen-Siersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotenburg-Fulda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saarbrücken
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schkeuditz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schwedt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuppertal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HumaPen Luxura | HumaPen Memoir
Started | 133 | 130
Received at Least One Dose of Study Drug | 131 | 130
Full Analysis Set (FAS) | 128 (Participants completed baseline and had at least 1 post-baseline measurement for efficacy analysis.) | 129 (Participants completed baseline and had at least 1 post-baseline measurement for efficacy analysis.)
Completed | 127 | 123
Not Completed | 6 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Sponsor decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HumaPen Luxura | HumaPen Memoir | Total
Number analyzed (Participants) | 128 | 129 | 257
Age Continuous [Mean (Standard Deviation); unit: years] | 41.2 (15.52) | 38.3 (17.37) | 39.8 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 56 | 108
  Male | 76 | 73 | 149
Race/Ethnicity, Customized [Number; unit: participants]
  White | 127 | 128 | 255
  Black or African American | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Germany | 128 | 129 | 257
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
  percentage of glycosylated hemoglobin | 9.06 (0.93) | 9.12 (1.04) | 9.09 (0.99)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24 Endpoint
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least Squares (LS) Mean values were controlled for treatment, visit, treatment*visit interaction, screening HbA1c (≤9% / >9%), change of prandial insulin at baseline, and baseline HbA1c.
Time Frame: Baseline, Week 24
Population: Participants in full analysis population set with missing values accounted for using mixed model repeated measures (MMRM).
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Arm/Group | HumaPen Luxura | HumaPen Memoir
Number analyzed (Participants) | 128 | 129
percentage of glycosylated hemoglobin | -0.48 [-0.64 to -0.32] | -0.43 [-0.59 to -0.28]
Statistical Analysis 1: Comparison: HumaPen Luxura vs HumaPen Memoir; Superiority criterion is met if the upper limit of Confidence Interval (CI) is below zero; Test type: Superiority or Other; p = 0.6692, Mixed Models Analysis; The model details are given in the section of Measure Description; LS Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.17 to 0.26], Standard Error of Mean 0.11

2. Secondary Outcome: Percentage of Participants Achieving Hemoglobin A1c (HbA1c) ≤7.5% and ≤7.0% at Week 24 Endpoint
Time Frame: Week 24
Population: Participants in full analysis population set who had Week 24 measurements.
Measure: Number; unit: percentage of participants
Arm/Group | HumaPen Luxura | HumaPen Memoir
Number analyzed (Participants) | 127 | 127
percentage of participants
  HbA1c ≤7.0% | 5.5 | 3.1
  HbA1c ≤7.5% | 16.5 | 11.0
Statistical Analysis 1: Comparison: HumaPen Luxura vs HumaPen Memoir; Test type: Superiority or Other; p = 0.3551, Chi-squared — P-value is for HbA1c ≤7.0%
Statistical Analysis 2: Comparison: HumaPen Luxura vs HumaPen Memoir; Test type: Superiority or Other; p = 0.2026, Chi-squared — P-value is for HbA1c ≤7.5%

3. Secondary Outcome: Score in Insulin Delivery System Questionnaire (IDSQ) - Willingness to Continue at Week 24 Endpoint
Description: IDSQ is used to evaluate acceptance of study pen. Willingness to continue was assessed by a single question, rated from 1 to 5 (1=Definitely unwilling and 5=Definitely willing). Higher score indicates stronger desire to continue. Least Squares (LS) Mean values were controlled for treatment and baseline score.
Time Frame: Week 24
Population: Participants in full analysis population set who had Week 24 measurements.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | HumaPen Luxura | HumaPen Memoir
Number analyzed (Participants) | 128 | 126
units on a scale | 4.06 [3.88 to 4.25] | 4.05 [3.86 to 4.23]
Statistical Analysis 1: Comparison: HumaPen Luxura vs HumaPen Memoir; Test type: Superiority or Other; p = 0.9070, ANCOVA; Analysis of covariance (ANCOVA) was adjusted for baseline values

4. Secondary Outcome: 30-Day Adjusted Rates of Self-Reported Hypoglycemic Episodes at Any Time From Baseline Through Week 24
Description: Hypoglycemic episode is defined as blood glucose measurement ≤3.9 millimoles/Liter (mmol/L; 70 milligrams/deciliter [mg/dL]). Adjusted rate = number of events in study period, divided by number of days in study period, then multiplied by 30.
Time Frame: Baseline through Week 24
Population: Randomized participants who took at least one dose of study drug with post-baseline hypoglycemia follow-up.
Measure: Mean (Standard Deviation); unit: number of events per 30 days
Arm/Group | HumaPen Luxura | HumaPen Memoir
Number analyzed (Participants) | 130 | 130
number of events per 30 days | 2.68 (4.66) | 2.46 (4.38)
Statistical Analysis 1: Comparison: HumaPen Luxura vs HumaPen Memoir; Test type: Superiority or Other; p = 0.9817, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: 30-Day Adjusted Rates of Self-Reported Hyperglycemic Episodes at Any Time From Baseline Through Week 24
Description: Hyperglycemic episode is defined as blood glucose measurement >18 mmol/L (324 mg/dL). Adjusted rate = number of events in study period, divided by number of days in study period, then multiplied by 30.
Time Frame: Baseline through Week 24
Population: Randomized participants who took at least one dose of study drug with post-baseline hyperglycemia follow-up.
Measure: Mean (Standard Deviation); unit: number of events per 30 days
Arm/Group | HumaPen Luxura | HumaPen Memoir
Number analyzed (Participants) | 130 | 130
number of events per 30 days | 2.56 (5.50) | 3.92 (9.82)
Statistical Analysis 1: Comparison: HumaPen Luxura vs HumaPen Memoir; Test type: Superiority or Other; p = 0.1187, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | HumaPen Luxura | HumaPen Memoir
Serious Adverse Events (participants affected / at risk) | 7/131 | 8/130
Other Adverse Events (participants affected / at risk) | 52/131 | 50/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HumaPen Luxura (N=131) | HumaPen Memoir (N=130)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HumaPen Luxura (N=131) | HumaPen Memoir (N=130)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (2)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (18) | 12 (13)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0)
Sinobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days